CLINICAL TRIAL: NCT07053202
Title: Clinical Study on TACE Combined With Immune Agents for Inhibiting Tumor Angiogenesis in Hepatocellular Carcinoma
Brief Title: TACE With Immune Agents for Angiogenesis in Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Wenhua Ma, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-B-035
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: TACE; Immune agents; Hepatic arterial infusion; Hepatocellular carcinoma; Tumor angiogenesis; Nivolumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE combined with Nivolumab (Experimental): Patients received TACE procedure. Additionally, hepatic artery infusion therapy with nivolumab was performed.
  Interventions: Combination Product: Nivolumab; Procedure: Transarterial Chemoembolization (TACE)
- TACE Alone (Active Comparator): Patients received TACE procedure alone.
  Interventions: Procedure: Transarterial Chemoembolization (TACE)

INTERVENTIONS:
Combination Product: Nivolumab — hepatic artery infusion therapy with nivolumab was performed
  Arms: TACE combined with Nivolumab
Procedure: Transarterial Chemoembolization (TACE) — Seldinger technique for femoral artery puncture. Catheterization to celiac trunk/hepatic artery. Infusion of a mixture of idarubicin, raltitrexed, iodized oil, and contrast agent (approx. 8 mL). Embolization with microspheres (300-500 μm and 500-700 μm).

SUMMARY:
This study investigates the clinical efficacy and safety of transarterial chemoembolization (TACE) combined with the immune agent nivolumab compared to TACE alone for treating hepatocellular carcinoma (HCC). The study aims to determine if the combination therapy can more effectively inhibit tumor angiogenesis, improve clinical benefit rates, and prolong survival, while maintaining a high safety profile.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common malignancy with high mortality. While TACE is a standard treatment, it can paradoxically stimulate tumor angiogenesis. Immune checkpoint inhibitors have shown promise in HCC, but single-agent efficacy is limited. This study was designed to evaluate whether combining TACE with hepatic arterial infusion of an immune agent (nivolumab) could improve outcomes by inhibiting tumor angiogenesis and enhancing anti-tumor immune responses. Patients diagnosed with unresectable HCC (BCLC stages A, B, C; Child-Pugh A or B) were randomized to receive either TACE alone (control group) or TACE combined with hepatic arterial infusion of nivolumab (study group). The study assessed objective response rate (ORR), disease control rate (DCR), changes in angiogenesis factors (VEGF, VEGFR-2, Ang-2) and tumor markers (CEA, AFP, CA199) before and one month after treatment. Adverse reactions, overall survival (OS), and progression-free survival (PFS) were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Diagnosis of HCC according to the Diagnosis and Treatment Guidelines for Primary Liver Cancer (2024 Edition), confirmed by pathological examination;
* Barcelona Clinic Liver Cancer (BCLC) stages A, B, and C, with non-resectable tumors;
* Liver function graded as Child-Pugh A or B;
* At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
* No severe hematologic abnormalities or immune deficiencies;
* Expected survival time >6 months.

Exclusion Criteria:

* Recurrent liver cancer or metastatic cancer from other organs;
* Previous treatment with other antitumor therapies, including surgery, radiotherapy, chemotherapy, targeted therapy, or immunotherapy;
* History of other malignant tumors;
* Pregnant or lactating women;
* Human immunodeficiency virus (HIV) infection;
* Severe cardiovascular, pulmonary, cerebral, or renal diseases;
* Active bleeding or coagulopathy outside the liver;
* Enrollment in another clinical trial or participation in a clinical trial within one month prior to admission;
* Psychiatric disorders or unstable mental status;
* Allergic reactions to the study drugs;
* Severe gastrointestinal diseases, such as active ulcers, or other conditions affecting drug absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Assessed at 1 month post-treatment, and then approximately every 3 months until disease progression, up to 24 months.
  Percentage of patients achieving Complete Remission (CR) or Partial Remission (PR) based on RECIST 1.1 criteria. ORR = [(CR + PR) / total cases] × 100%.
Disease Control Rate (DCR) | Assessed at 1 month post-treatment, and then approximately every 3 months until disease progression, up to 24 months.
  Percentage of patients achieving CR, PR, or Stable Disease (SD) based on RECIST 1.1 criteria. DCR = [(CR + PR + SD) / total cases] × 100%.

SECONDARY OUTCOMES:
Level of Vascular Endothelial Growth Factor (VEGF) | Baseline (one day before treatment) and 1 month after treatment.
  Serum level of Vascular Endothelial Growth Factor (VEGF) measured by ELISA.
Level of VEGF Receptor-2 (VEGFR-2) | Baseline (one day before treatment) and 1 month after treatment.
  Serum level of VEGF Receptor-2 (VEGFR-2) measured by ELISA.
Level of Angiopoietin-2 (Ang-2) | Baseline (one day before treatment) and 1 month after treatment.
  Serum level of Angiopoietin-2 (Ang-2) measured by ELISA.
Level of Carcinoembryonic Antigen (CEA) | Baseline (one day before treatment) and 1 month after treatment.
  Serum level of Carcinoembryonic Antigen (CEA) measured by ELISA.
Level of Alpha-fetoprotein (AFP) | Baseline (one day before treatment) and 1 month after treatment.
  Serum level of Alpha-fetoprotein (AFP) measured by ELISA.
Level of Carbohydrate Antigen 199 (CA199) | Baseline (one day before treatment) and 1 month after treatment.
  Serum level of Carbohydrate Antigen 199 (CA199) measured by ELISA.
Overall Survival (OS) | From randomization until death or end of study, whichever comes first, up to December 2023 (median follow-up 13.87 months).
  Time from randomization to death from any cause.
Progression-Free Survival (PFS) | From randomization until disease progression or death, whichever comes first, up to December 2023 (median follow-up 13.87 months).
  Time from randomization to disease progression (as per RECIST 1.1) or death from any cause.
Incidence of Adverse Reactions | From the first day of treatment until 30 days after the last treatment administration, monitored up to 24 months.
  Adverse reactions evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhua Ma, Principal Investigator — Department of Oncology, The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China